CLINICAL TRIAL: NCT05088070
Title: Phase I Clinical Study of SPH3348 Tablets, a C-Met Inhibitor, in Patients with Advanced Solid Tumors with C-Met Abnormalities
Brief Title: Clinical Study of SPH3348 Tablets, a C-Met Inhibitor, in Patients with Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Pharmaceuticals Holding Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPH3348-101
Record Dates: First submitted 2021-09-24; First posted 2021-10-21 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SPH 3348 tablets (Experimental): 6 different dosage group of SPH 3348 will be assigned with 16mg, 40mg, 80mg, 160mg, 240mg and 320mg respectively.
  Interventions: Drug: SPH 3348

INTERVENTIONS:
Drug: SPH 3348 — 2 tablets of 8mg SPH3348 will be orally administered once a day with empty stomach
Drug: SPH 3348 — 1 tablet of 40mg SPH3348 will be orally administered once a day with empty stomach
Drug: SPH 3348 — 2 tablets of 40mg SPH3348 will be orally administered once a day with empty stomach
Drug: SPH 3348 — 4 tablets of 40mg SPH3348 will be orally administered once a day with empty stomach
Drug: SPH 3348 — 6 tablets of 40mg SPH3348 will be orally administered once a day with empty stomach
Drug: SPH 3348 — 8 tablets of 40mg SPH3348 will be orally administered once a day with empty stomach

SUMMARY:
This is a phase 1 clinical trial of SPH3348 tablets, a c-Met inhibitor, in patients with advanced solid tumors with c-Met abnormalities. A modified 3 + 3 design was adopted in patients with advanced solid tumors with c-Met abnormalities, with a total of 6 dose groups, in which accelerated dose escalation was adopted for the lowest dose group, and 3 + 3 dose escalation was adopted from the second dose group. The primary objective was to evaluate the safety and tolerability of SPH3348 tablets in patients with advanced solid tumors with c-Met abnormalities.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced solid tumors with c-Met abnormalities who have failed standard of care or are not eligible for standard therapy currently
2. ECOG score of 0 or 1.
3. Patients must have measurable lesion that can be assessed by imaging per RECIST 1.1 criteria.
4. Expected survival > 12 weeks.
5. Patients must have adequate organ function
6. Patients must give informed consent to the study and sign the informed consent form prior to the trial.

Exclusion Criteria:

1. Received anti-tumor therapies, including but not limited to chemotherapy, biotherapy, radiotherapy, targeted therapy, etc., within 4 weeks prior to the first dose of study drug; received nitrosoureas or mitomycin C within 6 weeks prior to the start of study drug.
2. Received small molecule tyrosine kinase inhibitors within 2 weeks prior to the first dose.
3. Received strong CYP3A4 inducers or inhibitors or CYP3A4 substrates with narrow therapeutic windows within 2 weeks prior to the start of study drug.
4. Patients with active hepatitis B (hepatitis B surface antigen (HBsAg) positive) or hepatitis C (HCV).
5. Toxicities caused by prior treatments have not recovered to CTCAE Grade ≤ 1 or having ≥Grade 2 peripheral neuropathy, except for alopecia and other events judged as tolerable by the investigator.
6. Known allergy to any component of the reference drug.
7. Known drug or alcohol dependence.
8. Received surgical treatment including surgical and interventional procedures within 4 weeks prior to the start of study drug.
9. Patients with brain metastases.
10. Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment, or evidence of any clinically active interstitial lung disease.
11. Acute bacterial, viral, or fungal infection requiring systemic therapy or unexplained fever (temperature > 38.5 °C) during screening, prior to the first dose.
12. Neurological and psychiatric patients with obvious poor compliance.
13. Any of the following within 6 months prior to signing of informed consent form: uncontrolled congestive cardiac failure, severe or unstable angina pectoris, myocardial infarction, stroke, coronary/peripheral artery bypass surgery, pulmonary embolism.
14. Arrhythmia uncontrolled by medication or sustained QTcB prolongation.
15. Hypertension uncontrolled by medication
16. Participated in other drug clinical studies within 28 days prior to the first dose of study drug.
17. Women who are pregnant or in lactation period or women/men with childbearing plans.
18. Patients who cannot take oral medication, or have previous surgical history or serious gastrointestinal diseases such as dysphagia, active gastric ulcer, which may impair the absorption of the study drug in the investigator's opinion.
19. Other prior or current concomitant malignancies.
20. Patients who are ineligible to participate in this trial for any reason judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-07-02 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | 24 days
  Incidence of DLT in all subjects.
Maximum tolerated dose (MTD) | 24 days
  Measurement of MTD in all subjects.

SECONDARY OUTCOMES:
Maximum serum concentration (Cmax) of SPH 3348. | 24 days
  To characterize the PK (Pharmacokinetics) of SPH 3348.
Time of maximum serum concentration (Tmax) SPH 3348. | 24 days
  To characterize the PK (Pharmacokinetics) of SPH 3348.
Area under the concentration-time curve (AUC) of SPH 3348. | 24 days
  To characterize the PK (Pharmacokinetics) of SPH 3348.
Half-life (t1/2) of SPH 3348. | 24 days
  To characterize the PK (Pharmacokinetics) of SPH 3348.
Objective Response Rate (ORR) | 24 days
  Measurement of ORR in all subjects.
Disease control rate (DCR) | 24 days
  Measurement of DCR in all subjects.
Duration of remission (DOR) | 24 days
  Measurement of DOR in all subjects.
Progression-free survival (PFS) | 24 days
  Measurement of PFS in all subjects.
Biomarker expression level | 24 days
  Evaluate the level of hepatocyte growth factor(HGF).

CONTACTS AND LOCATIONS:
Overall Officials: Zishu Wang, Principal Investigator — The First Affliated Hospital of Bengbu Medical College; Huan Zhou, Principal Investigator — The First Affliated Hospital of Bengbu Medical College
Locations (1):
- The First Affliated Hospital of Bengbu Medical College, Bengbu, Anhui, China

IPD SHARING:
Plan to Share IPD: No